CLINICAL TRIAL: NCT06535048
Title: Effect of Fatty Liver on Antiviral Treatment in Patients With Hepatitis B
Brief Title: Impact of Fatty Liver on Hepatitis B Therapy
Acronym: AV-FLCHB
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AV-FLCHB; TJWJ2022XK034 (Other Grant/Funding Number: Tianjin Health Science and Technology Project key discipline special); TJYXZDXK-059B (Other Grant/Funding Number: Tianjin Key Medical Discipline (Specialty) Construction Project)
Record Dates: First submitted 2024-07-27; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Fatty Liver Disease; Chronic Hepatitis B; Antiviral Treatment
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fatty Liver: Hepatitis B patients with fatty liver
  Interventions: Drug: Entecavir；Tenofovir Disoproxil Fumarate (TDF)； Tenofovir alafenamide fumarate (TAF)；Interferons
- Non-Fatty Liver: Hepatitis B patients without fatty liver
  Interventions: Drug: Entecavir；Tenofovir Disoproxil Fumarate (TDF)； Tenofovir alafenamide fumarate (TAF)；Interferons

INTERVENTIONS:
Drug: Entecavir；Tenofovir Disoproxil Fumarate (TDF)； Tenofovir alafenamide fumarate (TAF)；Interferons — Entecavir: Participants will receive Entecavir 0.5 mg orally once daily for the duration of the study.
  Tenofovir Disoproxil Fumarate (TDF): Participants will receive TDF 300 mg orally once daily for the duration of the study.
  Tenofovir alafenamide fumarate (TAF): Participants will receive TAF 25 mg orally once daily for the duration of the study.
  Interferon (IFN): Participants will receive IFN 180 µg subcutaneously once weekly for at least 12 weeks.
  Other Names: Entecavir: Baraclude; Tenofovir Disoproxil Fumarate (TDF): Viread; Tenofovir Alafenamide Fumarate (TAF): Vemlidy; Pegylated Interferon Alpha (Peg-IFN-α): Pegasys

SUMMARY:
The primary goal of treating chronic hepatitis B(CHB) is to achieve maximal suppression of HBV replication, thereby reducing hepatocyte inflammation, necrosis, and liver fibrosis. Among various treatment strategies, antiviral therapy plays a crucial role. The prevalence of fatty liver disease (FLD) has continued to increase in recent decades. This study aims to accurately diagnose the pathological state of patients through liver biopsy and conduct a five-year follow-up to explore the impact of FLD on the efficacy of CHB treatment and to identify factors influencing adverse outcomes.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) remains a serious threat to people's health. As of 2019, approximately 296 million people (3.9% of the world's population) were infected with the HBV virus. In the treatment of CHB, Antiviral drugs can not only achieve long-term viral suppression for most CHB patients, but also have a positive impact on other CHB treatment goals and improvement of prognosis, but can not eliminate the risk of adverse clinical outcomes completely, which are partly attributed to concomitant diseases such as fatty liver disease (FLD). Both diseases can cause chronic liver injure and increase the risk of cirrhosis and HCC.All patients included in this study underwent liver biopsy to determine their pathological status, ensuring the reliability and accuracy of disease diagnosis. And based on biopsy results, patients were categorized into two groups:fatty liver combined with hepatitis B and hepatitis B alone. The main antiviral treatments used in the study include first-line NAs, such as entecavir, tenofovir disoproxil fumarate (TDF), tenofovir alafenamide fumarate (TAF), and interferons (IFN-α and Peg-IFN-α). They were followed for five years to thoroughly assess the long-term efficacy of antiviral treatment. Additionally, complications and liver fibrosis were evaluated using ultrasound and FibroScan to monitor the advancement of liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤75 years old, regardless of gender;
2. The patient had a positive hepatitis B marker and met the criteria for current hepatitis B virus infection (hepatitis B combined with fatty liver group);
3. Liver pathology indicated fatty liver (hepatitis B combined with fatty liver group);
4. All patients have complete medical history, B-ultrasound, FibroSan, hepatitis B five items, liver function and other laboratory test data.

Exclusion Criteria:

1. Aged <18 or >75 years old;
2. Patients diagnosed with or previously diagnosed with HCC;
3. Those who are co-infected with other hepatitis viruses (HAV, HCV, HDV, HEV) or HIV or syphilis;
4. The follow-up data of patients are seriously missing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients between the ages of 18 and 75 who underwent liver biopsies and were diagnosed with chronic hepatitis B (CHB), all of whom received antiviral therapy for the first time. Patients were divided into two groups according to whether they had fatty liver. All patients had a complete history, including B-ultrasound, fiber scan, hepatitis B serology, liver function tests and other examination data.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of virological levels in serum | 5 years
  The incidence of negativity for HBV DNA, HBsAg, and HBeAg, defined as serum levels less than 20 IU/mL, 0.05 IU/mL, and 1.0 S/CO, respectively.
Comparison of liver function improvement | 5 years
  Liver function was assessed by measuring serum ALT, AST, and GGT levels during treatment.

SECONDARY OUTCOMES:
Impact of Fatty Liver on the Incidence of Adverse Outcomes in CHB Patients | 5 years
  Evaluation of the incidence of adverse outcomes such as liver cirrhosis, hepatocellular carcinoma (HCC) under ultrasound, and overall survival in CHB patients with fatty liver compared to those without fatty liver.
Factors affecting adverse outcomes in patients with chronic hepatitis B | 5 years
  Kaplan-Meier method was used for survival analysis, and the influencing factors of poor prognosis were analyzed.

IPD SHARING:
Plan to Share IPD: No
Due to concerns about participant privacy, data security, and the administrative burden of managing data requests, individual participant data (IPD) will not be shared. Additionally, the current research agreement does not include a data sharing clause.